CLINICAL TRIAL: NCT02853825
Title: Randomized Controlled Trial of the Jewish Family & Children's Service of the Suncoast, Inc.'s Healthy Families/Healthy Children Program
Brief Title: RCT of the Jewish Family & Children's Services (JFCS) HFHC Program
Acronym: JFCS:HFHC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jewish Family & Children's Service of the Suncoast, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016/06/35; 90FM0070 (Other Grant/Funding Number: HHS, ACF, Office of Family Assistance)
Record Dates: First submitted 2016-07-28; First posted 2016-08-03 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Family Relations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait List Control Group (No Intervention): No interventions given, this is a wait list control group.
- Intervention Group (Experimental): Receive relationship skill enhancement classes with access to parenting, employment services, and financial services.
  Interventions: Behavioral: Relationship Skill Enhancement

INTERVENTIONS:
Behavioral: Relationship Skill Enhancement — Receive relationship classes with access to parenting, employment services, and financial services.
  Arms: Intervention Group

SUMMARY:
Every program element was designed to ensure that all children in the areas served will live in stable, happy, healthy family situations. The JFCS Healthy Families/Healthy Children program will provide relationship skill enhancement interventions. All program participants in the intervention group will have acces to: parenting skill enhancement interventions, employment readiness and/or situation enhancement, as well as financial knowledge and/or situation enhancement.

DETAILED DESCRIPTION:
The goal of the Healthy Families/Healthy Children (HFHC) program is to ensure that all children in The Region live in stable, happy, healthy family situations. HFHC will be able to deliver existing services that have proven effective and new services that are research-based. Need to be addressed: Unhealthy relationships, inadequate parental skills and attitudes related to nurturing and responsible parenting, lack of knowledge of finances and/or economic self sufficiency, underdeveloped employment readiness skills, difficult-to-access job opportunities and housing. Proposed Services: In conjunction with a wide-range of community partners operating a comprehensive system of care, JFCS will provide a public advertising campaign, Marriage and Relationship Education/Skills (MRES), Nurturing Parenting education, financial management education and services, and job career advancement services. HFHC is designed around a strong marriage and relationship education/skills (MRES) component. The program includes parenting skills classes, a robust effort to address participation barriers, and partnership with local employment and employment skill-building agencies to address the economic stability needs of participants. Case management and support service coordination ensure comprehensive service delivery for every participant. Participants will have meaningful improvements in marriage/relationship skills, improved parenting/co-parenting skills, improved family functioning,improved adult and child well-being, and increased economic stability/reduced poverty. Population groups to be served: Low-income individuals, couples, engaged couples, and married couples 18 years of age up to 64 years of age and their family members.Research component: The project will conduct a randomized controlled trial to test hypotheses regarding our program's effectiveness. The Control group will be on a wait list and will not receive the Intervention (i.e., program services) until their final post-test measures are completed.

ELIGIBILITY:
Inclusion Criteria:

* Residents of Sarasota and Manatee Counties

Exclusion Criteria:

* No minors
* No one over 64 years of age

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 786 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
The Family Environment Scale | 26 Weeks
Dyadic Adjustment Scale | 26 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Young, PhD, Principal Investigator — Jewish Family & Children's Services
Locations (1):
- JFCS, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: No